CLINICAL TRIAL: NCT03440489
Title: Assessment of Skeletal Muscle Dysfunction in Patient With Idiopathic Pulmonary Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, seham abd elmouty, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SMD
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Interstitial Lung Disease; Skeletal Muscle Dysfunction
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: skeletal muscle dysfunction in patient with idiopathic pulmonary fibrosis six minute walking test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- six-minute walking test (Other): physical performance of the muscle: measured by Gait speed test, Timed up and go test, six-minute walking test , 30 seconds chair stand test
  Interventions: Diagnostic Test: Six-minute walking test; Diagnostic Test: 30 seconds chair stand test

INTERVENTIONS:
Diagnostic Test: Six-minute walking test — physical performance of the muscle measured by these tests
  Other Names: Gait speed test; Timed up and go test
Diagnostic Test: 30 seconds chair stand test — physical performance of the muscle measured by these tests

SUMMARY:
Interstitial lung disease includes a heterogeneous group of chronic lung conditions that is characterized by exertional dyspnoea and poor health related quality of life . includes idiopathic pulmonary fibrosis of unknown cause And another groups are caused by occupational, inorganic or organic exposure, drug- induced toxicities, or are secondaries to connective tissue disease The clinical course and outcome of interstitial lung diseases are highly variable between different sub types, but survival after diagnosis of idiopathic pulmonary fibrosis is only 2.5 to 5 years is a progressive and fibrosing lung disease that is characterized by architectural distortion of the lung parenchyma and is progressive, with a dismal prognosis Also patient with idiopathic pulmonary fibrosis generally demonstrate greater abnormalities of exercise induced gas exchange than those with other forms of Interstitial lung disease

DETAILED DESCRIPTION:
Interstitial lung disease includes a heterogeneous group of chronic lung conditions that is characterized by exertional dyspnoea and poor health related quality of life . includes idiopathic pulmonary fibrosis of unknown cause And another groups are caused by occupational, inorganic or organic exposure, drug- induced toxicities, or are secondaries to connective tissue disease The clinical course and outcome of interstitial lung diseases are highly variable between different sub types, but survival after diagnosis of idiopathic pulmonary fibrosis is only 2.5 to 5 years is a progressive and fibrosing lung disease that is characterized by architectural distortion of the lung parenchyma and is progressive, with a dismal prognosis Also patient with idiopathic pulmonary fibrosis generally demonstrate greater abnormalities of exercise induced gas exchange than those with other forms of Interstitial lung disease People with exhibit limitation in peak exercise capacity, which is associated with impaired ventilation, gas exchange and pulmonary perfusion abnormalities Also in people with interstitial lung diseases there is a relationship between quadriceps muscle weakness and exercise capacity raising the importance of skeletal muscle dysfunction. Furthermore, since interstitial lung diseases is the leading diagnosis referred for lung transplant characterizing skeletal muscle dysfunction and its relationship to exercise capacity prior to lung transplant is of specific interest for this population.

The cause of muscle dysfunction in individuals with lung disease is multifactorial, including factors such as disuse, hypoxaemia, malnutrition, oxidative stress, systemic inflammation and medication Pulmonary inflammation and oxidative stress are thought to be pivotal in the pathogenesis of idiopathic interstitial pneumonia

ELIGIBILITY:
Inclusion Criteria:

* All patient who will be presented to assuit chest department and diagnosed as IPF.

Exclusion Criteria:

* 1-IPF patient with malignant tumors. 2-Comorbid end stage renal, cardiac or hepatic patient. 3-patient who refused to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
assess skeletal muscle dysfunction in interstitial lung diseased patients by 30 seconds chair stand test | 30 seconds
  30 seconds chair stand test

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd El-ghany, Study Chair — Assiut University; Atef el karn, Study Chair — Assiut University; Sahar Farghaly yuessif, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Collard HR, King TE Jr, Bartelson BB, Vourlekis JS, Schwarz MI, Brown KK. Changes in clinical and physiologic variables predict survival in idiopathic pulmonary fibrosis. Am J Respir Crit Care Med. 2003 Sep 1;168(5):538-42. doi: 10.1164/rccm.200211-1311OC. Epub 2003 May 28. PMID 12773325
- [Background] Travis WD, Costabel U, Hansell DM, King TE Jr, Lynch DA, Nicholson AG, Ryerson CJ, Ryu JH, Selman M, Wells AU, Behr J, Bouros D, Brown KK, Colby TV, Collard HR, Cordeiro CR, Cottin V, Crestani B, Drent M, Dudden RF, Egan J, Flaherty K, Hogaboam C, Inoue Y, Johkoh T, Kim DS, Kitaichi M, Loyd J, Martinez FJ, Myers J, Protzko S, Raghu G, Richeldi L, Sverzellati N, Swigris J, Valeyre D; ATS/ERS Committee on Idiopathic Interstitial Pneumonias. An official American Thoracic Society/European Respiratory Society statement: Update of the international multidisciplinary classification of the idiopathic interstitial pneumonias. Am J Respir Crit Care Med. 2013 Sep 15;188(6):733-48. doi: 10.1164/rccm.201308-1483ST. PMID 24032382